CLINICAL TRIAL: NCT05387083
Title: A Phase 2a, Randomized, Double-Blind, Placebo Controlled, Single-Center, Human Tick Kill Proof-of-Concept Study Evaluating the Safety, Tolerability, and Whole Blood Concentration of TP-05 (lotilaner) in Healthy Volunteers
Brief Title: A Human Tick Kill Study to Investigate the Safety, Tolerability, and Whole Blood Concentration of TP-05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: TRS-015
Record Dates: First submitted 2022-05-03; First posted 2022-05-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteer
Keywords: Lyme Disease; Ticks
MeSH Terms: conditions — Lyme Disease | interventions — lotilaner

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose of TP-05 (lotilaner) (Experimental): Single Oral Low Dose of TP-05 tablet.
  Interventions: Drug: Low Dose TP-05
- High Dose of TP-05 (lotilaner) (Experimental): Single Oral High Dose of TP-05 tablet.
  Interventions: Drug: High Dose TP-05
- Placebo (Placebo Comparator): Single Oral Dose of placebo tablet.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Low Dose TP-05 — Healthy Volunteers will receive a single low dose of TP-05 on Day 1.
  Other Names: Lotilaner
  Arms: Low Dose of TP-05 (lotilaner)
Drug: High Dose TP-05 — Healthy Volunteers will receive a single high dose of TP-05 on Day 1.
  Other Names: Lotilaner
  Arms: High Dose of TP-05 (lotilaner)
Drug: Placebo Comparator — Healthy Volunteers will receive a single dose of placebo on Day 1.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2a, randomized, double-blind, proof-of-concept, single-center study evaluating the safety, tolerability, and whole blood concentration of TP-05 (lotilaner) in the killing of ticks after they have attached to human skin.

DETAILED DESCRIPTION:
The study will consist of a screening period of no more than 30 days. Participants will come to the study center on Day -1 for tick placements on the skin. Nymphal ticks that have been tested negative for human pathogens and are known to be ready to attach will be placed.

On Day 1, the number of attached, live ticks will be counted. Participants will be randomized on Day 1 to receive either low dose or high dose of TP-05 or placebo. Tick attachment and mortality will be completed on Day 1 and after participants' return to the study center on Day 2 (24 hours after dosing). Participants will have ticks removed from the skin at the study center after the Day 2 (24 hours) tick count.

Participants will come to the study center on Day 30 for another placement of ticks on the skin. Tick attachment and mortality will be determined on Day 30 and on Day 31 (24 hours after placement).

Participants will complete the treatment period at Day 60. Participants will undergo a long-term safety follow-up period which will include additional safety and PK visits through Day 301.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 to 59 years of age inclusive, at the time of signing the informed consent.
2. Participants who are overtly healthy as determined by medical evaluation including having no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination.
3. Participants who are non- or ex-smokers.
4. Willingness to comply with all study procedures and availability for the duration of the study.
5. BMI within the range 18 - 32 kg/m2
6. Willingness to comply with contraceptive requirements
7. Capable of giving signed informed consent

Exclusion Criteria:

1. Female who is lactating at Screening.
2. Female who is pregnant according to the serum pregnancy test at Screening or prior to study treatment administration.
3. History of significant hypersensitivity to lotilaner or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
4. Presence or history of significant gastrointestinal, metabolic, liver or kidney disease, or surgery that may affect drug bioavailability (excluding appendectomy).
5. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease.
6. Have a history of malignancy (or active malignancy), with the exception of treated basal cell or squamous cell carcinoma.
7. Presence of clinically significant ECG abnormalities at Screening, as defined by the Investigator.
8. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse.
9. Any clinically significant illness in the 28 days prior to study treatment administration.
10. Known history of chronic infectious disease.
11. History of allergy to surgical tape, hydrocolloid, or dressing.
12. History of severe reactions to tick bites (granuloma or systemic reactions).
13. Use of any non-prescription or prescription drugs (with the exception of hormonal contraceptives, hormone replacement therapy, acetaminophen) in the 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to study treatment administration.
14. Use of St. John's wort in the 28 days prior to study treatment administration.
15. Intake of lotilaner in the 6 months prior to study treatment administration.
16. Treatment with an investigational drug within 30 days or 5 times the half-life (whichever is longer) prior to Screening.
17. History of live attenuated vaccine within 4 weeks prior to randomization or requirement to receive these vaccinations at any time during the study.
18. Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of the Investigator, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data.
19. Blood donation of approximately 500 mL within 56 days prior to Screening.
20. Plasma donation within 7 days prior to Screening.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
The Incidence of treatment emergent adverse events from baseline | Day -1 through Day 301
  Safety and tolerability will be evaluated by incidence rate of treatment emergent adverse events from baseline.
Clinically significant changes from Baseline chemistry laboratory tests | Day -1 through Day 301
  Number of participants with clinically significant changes in clinical laboratory tests
Clinically significant changes from Baseline hematology laboratory tests | Day -1 through Day 301
  Number of participants with clinically significant changes in clinical laboratory tests
Clinically significant changes from Baseline vital signs | Day -1 through Day 301
  Number of participants with clinically significant changes in vital signs.
Clinically significant changes from Baseline electrocardiograms (ECGs) | Day -1 through Day 301
  Safety will be assessed by evaluating clinically significant changes from Baseline ECGs change in mean ventricular rate [beats/min]
Clinically significant changes from Baseline electrocardiograms (ECGs) measures | Day -1 through Day 301
  Safety will be assessed by evaluating clinically significant changes from Baseline ECGs change in pulse rate [msec]
Clinically significant changes from Baseline QTC interval | Day -1 through Day 301
  Safety will be assessed by evaluating clinically significant changes from Baseline ECGs change in QTC interval
Clinically significant changes from Baseline QRS interval | Day -1 through Day 301
  Safety will be assessed by evaluating clinically significant changes from Baseline ECGs change in QRS interval

SECONDARY OUTCOMES:
Evaluate the concentration of lotilaner in whole blood | Day -1 through Day 301
  Measure of concentration of lotilaner in whole blood at specified timepoints
TP-05 on Tick Mortality | Day 2 through Day 31
  Evaluate Tick Mortality after TP-05 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Dhamdhere, MD, PhD, Study Director — Tarsus Pharmaceuticals, Inc.; Linden Hu, MD, Principal Investigator — Tufts University School of Medicine; Yoav Golan, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts University School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No